CLINICAL TRIAL: NCT01504321
Title: Polycystic Ovary Syndrome - Targeting the Sympathetic Nervous System to Improve Outcomes
Brief Title: Polycystic Ovary Syndrome - Improving Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Principal Investigator, Markus Schlaich, Associate Professor, Baker Heart and Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Human Neuro -PCOS
Record Dates: First submitted 2012-01-02; First posted 2012-01-05 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary syndrome; PCOS; sympathetic nervous system; moxonidine
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — moxonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Active (Active Comparator)
  Interventions: Drug: Moxonidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxonidine — 0.2 mg/day moxonidine for 2 weeks 0.4 mg/day moxonidine for 3 months
  Arms: Active
Drug: Placebo — Encapsulated lactose powder
  Arms: Placebo

SUMMARY:
Polycystic ovary syndrome affects a striking 9-18% of Australian reproductive aged women and has been associated with a number of metabolic abnormalities.

Given the strong correlation between metabolic abnormalities and increased sympathetic activity, we hypothesise that reducing this activity using medication (moxonidine) can help improve the metabolic abnormalities, and therefore improve outcomes in polycystic ovary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and class I obese pre-menopausal women
* Diagnosis of PCOS by Rotterdam criteria

Exclusion Criteria:

* Any current medication
* pregnancy or the desire to become pregnant
* BMI > 35
* a history of type I diabetes, secondary hypertension not due to PCOS
* cardiovascular, cerebrovascular, liver or thyroid disease
* severe mental illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Microneurography | 3 months
  Microneurography is a technique developed to measure the sympathetic activitiy directly from the peroneal nerve. Microneurography will be performed at baseline visit and at 3 months follow up visit.

SECONDARY OUTCOMES:
Blood biochemistry measurement | 3 months
  To assess the metabolic function of the participants we will be drawing fasting blood samples for biochemical analysis. These test will be performed at baseline and 3 months follow up visit
Oral glucose tolerance test | 3 months
  A standard 75g glucose tolerance test will be performed. Venous blood will be taken before and 2 hours after the glucose drink was given.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Lambert, Dr, Principal Investigator — BakerIDI Heart and Diabetes Institute
Locations (1):
- Heart Centre, Alfred Hospital, Prahran, Victoria, Australia

REFERENCES:
- [Derived] Jewson J, Lambert E, Sari C, Jona E, Shorakae S, Lambert G, Gaida J. Does moxonidine reduce Achilles tendon or musculoskeletal pain in women with polycystic ovarian syndrome? A secondary analysis of a randomised controlled trial. BMC Endocr Disord. 2020 Aug 26;20(1):131. doi: 10.1186/s12902-020-00610-8. PMID 32847570
- [Derived] Shorakae S, Jona E, de Courten B, Lambert GW, Lambert EA, Phillips SE, Clarke IJ, Teede HJ, Henry BA. Brown adipose tissue thermogenesis in polycystic ovary syndrome. Clin Endocrinol (Oxf). 2019 Mar;90(3):425-432. doi: 10.1111/cen.13913. Epub 2019 Jan 7. PMID 30548504
- [Derived] Shorakae S, Lambert EA, Jona E, Ika Sari C, de Courten B, Dixon JB, Lambert GW, Teede HJ. Effect of Central Sympathoinhibition With Moxonidine on Sympathetic Nervous Activity in Polycystic Ovary Syndrome-A Randomized Controlled Trial. Front Physiol. 2018 Oct 25;9:1486. doi: 10.3389/fphys.2018.01486. eCollection 2018. PMID 30410448